CLINICAL TRIAL: NCT00377611
Title: A Study to Investigate the Incidence of Influenza and Influenza-related Complications, in Adults Between 50-64 Years and Elderly Adults 65 Years and Over Vaccinated With Fluarix™
Brief Title: Study on the Incidence of Influenza and Its Complications, in Subjects Aged 50 Years and Over Vaccinated With Fluarix™
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 107564
Record Dates: First submitted 2006-09-15; First posted 2006-09-18 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-06

CONDITIONS: Influenza
Keywords: Influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (2):
- FLUARIX 50-64 YEARS GROUP (Experimental): Adult subjects aged between and including 50-64 years who received a single dose of Fluarix™ vaccine intramuscularly into the deltoid region of the non-dominant arm, were enrolled for investigation of influenza and influenza-related complications.
  Interventions: Biological: Fluarix™
- FLUARIX 65+ YEARS GROUP (Experimental): Elderly subjects aged 65 and over who received a single dose of Fluarix™ vaccine intramuscularly into the deltoid region of the non-dominant arm, were enrolled for investigation of influenza and influenza-related complications.
  Interventions: Biological: Fluarix™

INTERVENTIONS:
Biological: Fluarix™

SUMMARY:
A study to investigate the incidence of influenza and influenza-related complications, in adults between 50-64 years and elderly adults 65 years and over vaccinated with Fluarix™

ELIGIBILITY:
Inclusion Criteria:

* A male or female age 50 years or older at the time of the first vaccination.
* non-childbearing female
* Availability to follow up by phone
* Subjects with residence status allowing free mixing with general community

Exclusion Criteria:

* Use of non-registered products
* Pregnancy
* Hypersensitivity to a previous dose of influenza vaccine
* Acute disease at the time of enrolment/vaccination.
* History of allergy or reactions likely to be exacerbated by any component of the vaccine
* Any contra-indication to intramuscular administration of Fluarix™
* For subjects enrolled in the immunogenicity subset only: administration of immune-modifying drugs within 7 days prior to the vaccination

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3054 (Actual)
Dates: Start 2006-10-05 (Actual); Primary Completion 2007-06-20 (Actual); Study Completion 2007-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (31):
- United States (9):
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Delray Beach, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Somers Point, New Jersey
  - GSK Investigational Site, Camillus, New York
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Norfolk, Virginia
- Germany (15):
  - GSK Investigational Site, Güglingen, Baden-Wurttemberg
  - GSK Investigational Site, Rudersberg, Baden-Wurttemberg
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Rhaunen, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- GSK Investigational Site, Utrecht, Netherlands
- Poland (6):
  - GSK Investigational Site, Dębica
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Mielec
  - GSK Investigational Site, Porąbka
  - GSK Investigational Site, Siemianowice Śląskie
  - GSK Investigational Site, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 107564 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 107564 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107564 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107564 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 107564 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107564 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluarix 50-64 Years Group | Fluarix 65+ Years Group
Started | 1047 | 2007
Completed | 1025 | 1974
Not Completed | 22 | 33
Not completed — Adverse Event | 2 | 9
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 0 | 5
Not completed — Lost to Follow-up | 18 | 16
Not completed — Other | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluarix 50-64 Years Group | Fluarix 65+ Years Group | Total
Number analyzed (Participants) | 1047 | 2007 | 3054
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.6 (4.11) | 70.3 (4.42) | 65.92 (7.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 599 | 1094 | 1693
  Male | 448 | 913 | 1361

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With at Least One Influenza-like-infection (ILI) Episode
Description: Analysis included all non-confirmed or lab confirmed ILI episodes (at least 1 episode, 1 episode, 2 episodes or more than (>) 2 episodes) reported.
Time Frame: From Month 0 to Month 6
Population: The analysis was performed on the Total Vaccinated Cohort which included all subjects with one vaccine administration documented, for whom data were available.
Measure: Count of Participants; unit: Participants
Groups:
- Fluarix 50+ Years Group: Adult subjects aged 50 and over who received a single dose of Fluarix™ vaccine intramuscularly into the deltoid region of the non-dominant arm, were enrolled for investigation of influenza and influenza-related complications.
Arm/Group | Fluarix 50-64 Years Group | Fluarix 65+ Years Group | Fluarix 50+ Years Group
Number analyzed (Participants) | 297 | 697 | 994
Participants
  At least 1 ILI episode | 133 | 243 | 376
  1 ILI episode | 125 | 231 | 356
  2 ILI episodes | 8 | 12 | 20
  >2 ILI episodes | 0 | 0 | 0

2. Primary Outcome: Number of Subjects With Laboratory-confirmed Influenza Infection Type A and/or Type B
Description: Lab confirmed ILI episodes were assessed by means of viral culture (VC) infection (nasal and throat swabs) determination and/or using the Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) assay.
Time Frame: From Month 0 to Month 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 50-64 Years Group | Fluarix 65+ Years Group | Fluarix 50+ Years Group
Number analyzed (Participants) | 297 | 697 | 994
Participants
  VC and/or RT-PCR Influenza A and/or B | 13 | 15 | 28
  VC and/or RT-PCR Influenza A | 13 | 15 | 28
  VC and/or RT-PCR Influenza B | 0 | 0 | 0
  VC and/or RT-PCR Influenza A and B | 0 | 0 | 0
  VC Influenza A and/or B | 12 | 9 | 21
  VC Influenza A | 12 | 9 | 21
  VC Influenza B | 0 | 0 | 0
  VC Influenza A and B | 0 | 0 | 0
  RT-PCR Influenza A and/or B | 13 | 15 | 28
  RT-PCR Influenza A | 13 | 15 | 28
  RT-PCR Influenza B | 0 | 0 | 0
  RT-PCR Influenza A and B | 0 | 0 | 0
  VC and RT-PCR Influenza A and/or B | 12 | 9 | 21
  VC and RT-PCR Influenza A | 12 | 9 | 21
  VC and RT-PCR Influenza B | 0 | 0 | 0
  VC and RT-PCR Influenza A and B | 0 | 0 | 0

3. Primary Outcome: Number of Subjects With Hospitalization, Emergency Room Visits, or Unscheduled Medical Office Visits Due to ILI
Description: ILI which led to subject hospitalization, emergency room visits and unplanned medical office visits were recorded by number (at least 1, 1, or above 1), as part of the ILI surveillance.
Time Frame: From Month 0 to Month 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 50-64 Years Group | Fluarix 65+ Years Group | Fluarix 50+ Years Group
Number analyzed (Participants) | 297 | 697 | 994
Participants
  At least 1 ILI | 31 | 51 | 82
  1 ILI | 31 | 49 | 80
  Above 1 ILI | 0 | 2 | 2

4. Primary Outcome: Number of Subjects With Hospitalizations, Emergency Room Visits or Unscheduled Medical Office Visits, Due to Laboratory Confirmed Influenza
Description: Laboratory confirmed (LC) ILI which led to subject hospitalization, emergency room visits and unplanned medical office visits were recorded by number (at least 1, 1, or above 1), as part of the ILI surveillance.
Time Frame: From Month 0 to Month 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 50-64 Years Group | Fluarix 65+ Years Group | Fluarix 50+ Years Group
Number analyzed (Participants) | 297 | 697 | 994
Participants
  At lesat 1 LC ILI | 2 | 6 | 8
  1 LC ILI | 2 | 6 | 8
  Above 1 LC ILI | 0 | 0 | 0

5. Primary Outcome: Number of Subjects With Hospitalization or Emergency Room Visit for Any Cause
Description: As part of ILI surveillance any reasons, or other reasons than those mentioned which led to subject hospitalization, emergency room visits and unplanned medical office visits were recorded by number (at least 1, 1, or above 1).
Time Frame: From Month 0 to Month 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 50-64 Years Group | Fluarix 65+ Years Group | Fluarix 50+ Years Group
Number analyzed (Participants) | 297 | 697 | 994
Participants
  Any reason - at least 1 | 47 | 124 | 171
  Any reason - one | 43 | 107 | 150
  Any reason - above one | 4 | 17 | 21
  Other reason - at least 1 | 13 | 72 | 85
  Other reason - one | 10 | 69 | 79
  Other reason - above 1 | 3 | 3 | 6

6. Primary Outcome: Number of Subjects With Emergency Room Visits, or Unscheduled Medical Office Visits Due to Influenza-related Complications
Description: ILI complications which led to subject hospitalization, emergency room visits and unplanned medical office visits were recorded by number (at least 1, 1, or above 1) as part of the ILI surveillance, which included: pneumonia, ischemic heart disease, congestive failure, acute cerebrovascular disease chronic obstructive pulmonary disease (COPD) exacerbation.
Time Frame: From Month 0 to Month 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 50-64 Years Group | Fluarix 65+ Years Group | Fluarix 50+ Years Group
Number analyzed (Participants) | 297 | 697 | 994
Participants
  At least 1 ILI complication | 4 | 16 | 20
  1 ILI complication | 4 | 14 | 18
  Above 1 ILI complication | 0 | 2 | 2

7. Primary Outcome: Number of Subjects With Influenza-related Complications
Description: ILI complications refer to episodes of pneumonia, ischemic heart disease [HD] (unstable angina or myocardial infarction), congestive heart failure [HF], acute cerebrovascular disease [ACD] (stroke or transient ischemic attack [IA]), COPD exacerbation and all illnesses (pooled episode of each illness). ILI complications were recorded by number of episodes (at least 1 episode, 1 episode and above 1 episode).
Time Frame: From Month 0 to Month 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 50-64 Years Group | Fluarix 65+ Years Group | Fluarix 50+ Years Group
Number analyzed (Participants) | 297 | 697 | 994
Participants
  Pneumonia at least 1 episode | 2 | 9 | 11
  Pneumonia 1 episode | 2 | 9 | 11
  Pneumonia above 1 episode | 0 | 0 | 0
  Ischemic HD at least 1 episode | 2 | 3 | 5
  Ischemic HD 1 episode | 2 | 3 | 5
  Ischemic HD above 1 episode | 0 | 0 | 0
  Unstable angina at least 1 episode | 0 | 0 | 0
  Unstable angina 1 episode | 0 | 0 | 0
  Unstable angina above 1 episode | 0 | 0 | 0
  Myocardial infarction at least 1 episode | 2 | 3 | 5
  Myocardial infarction 1 episode | 2 | 3 | 5
  Myocardial infarction above 1 episode | 0 | 0 | 0
  Congestive HF at least 1 episode | 0 | 2 | 2
  Congestive HF 1 episode | 0 | 2 | 2
  Congestive HF above 1 episode | 0 | 0 | 0
  ACD at least 1 episode | 0 | 1 | 1
  ACD 1 episode | 0 | 1 | 1
  ACD above 1 episode | 0 | 0 | 0
  Stroke at least 1 episode | 0 | 1 | 1
  Stroke 1 episode | 0 | 1 | 1
  Stroke above 1 episode | 0 | 0 | 0
  Transient IA at least 1 episode | 0 | 0 | 0
  Transient IA 1 episode | 0 | 0 | 0
  Transient IA above 1 episode | 0 | 0 | 0
  COPD exacerbation at least 1 episode | 1 | 3 | 4
  COPD exacerbation 1 episode | 1 | 2 | 3
  COPD exacerbation above 1 episode | 0 | 1 | 1
  Any illness at least 1 episode | 5 | 17 | 22
  Any illness 1 episode | 5 | 15 | 20
  Any illness above 1 episode | 0 | 2 | 2

8. Primary Outcome: Number of Subjects With Fatal Outcomes Due to Laboratory Confirmed Influenza Infection
Description: Death due to lab confirmed influenza infection was recorded during the influeza period only.
Time Frame: From Month 0 to Month 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 50-64 Years Group | Fluarix 65+ Years Group | Fluarix 50+ Years Group
Number analyzed (Participants) | 1047 | 2007 | 3054
Participants | 0 | 0 | 0

9. Primary Outcome: Number of Subjects With Fatal Outcomes
Description: Number of deaths caused by laboratory non-confirmed ILI or other reasons were recorded during the influenza
Time Frame: From Month 0 to Month 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 50-64 Years Group | Fluarix 65+ Years Group | Fluarix 50+ Years Group
Number analyzed (Participants) | 1047 | 2007 | 3054
Participants
  ILI not confirmed | 0 | 0 | 0
  Other | 1 | 6 | 7

10. Primary Outcome: Number of Subjects With Laboratory-confirmed Respiratory Syncytial Virus Infection (RSV)
Description: RSV infection was determined by the RT-PCR assay.
Time Frame: From Month 0 to Month 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 50-64 Years Group | Fluarix 65+ Years Group | Fluarix 50+ Years Group
Number analyzed (Participants) | 297 | 697 | 994
Participants | 16 | 27 | 43

11. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination and related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: From Month 0 to Month 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 50-64 Years Group | Fluarix 65+ Years Group | Fluarix 50+ Years Group
Number analyzed (Participants) | 1047 | 2007 | 3054
Participants | 23 | 105 | 128

12. Primary Outcome: Number of Seroconverted Subjects for Each Influenza Strain
Description: A seroconverted subject was defined as a subject having either a pre-vaccination hemagglutinin inhibition (HI) titer lower than (<) 1:10 and a post-vaccination titer greater than or equal to (≥) 1:40, or a pre-vaccination titer ≥1:10 and a minimum four-fold increase in the post-vaccination titer. Assessed influenza strains were A/New Caledonia, A/Wisconsin and B/Malaysia.
Time Frame: At Day 21
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects for whom data concerning immunogenicity measures were available. This included subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 50-64 Years Group | Fluarix 65+ Years Group | Fluarix 50+ Years Group
Number analyzed (Participants) | 171 | 307 | 478
Participants
  A/New Caledonia | 171 | 306 | 477
  A/Wisconsin | 167 | 304 | 471
  B/Malaysia | 168 | 306 | 474

13. Primary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against 3 Strains of Influenza Disease
Description: The seroconversion factor (SCF) was defined as the fold increase in serum HI geometric mean titer (GMT) post vaccination on Day 21 compared to Day 0. The 3 influenza strains assessed were A/New Caledonia, A/Wisconsin and B/Malaysia.
Time Frame: At Day 21
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Fluarix 50-64 Years Group | Fluarix 65+ Years Group | Fluarix 50+ Years Group
Number analyzed (Participants) | 171 | 307 | 478
Titer
  A/New Caledonia | 216.4 [180.8 to 259.0] | 142.9 [125.8 to 162.4] | 165.8 [149.2 to 184.2]
  A/Wisconsin | 156.7 [125.3 to 196.0] | 179.1 [154.0 to 208.4] | 170.8 [150.6 to 193.6]
  B/Malaysia | 149.9 [124.3 to 180.9] | 184.0 [161.9 to 209.2] | 171.0 [153.8 to 190.2]

14. Primary Outcome: Number of Seroprotected Subjects Against the 3 Influenza Strains
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer ≥1:40.
Time Frame: At Day 0 (PRE)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 50-64 Years Group | Fluarix 65+ Years Group | Fluarix 50+ Years Group
Number analyzed (Participants) | 171 | 307 | 478
Participants
  A/New Caledonia, PRE | 91 | 184 | 275
  A/Wisconsin, PRE | 48 | 106 | 154
  B/Malaysia, PRE | 63 | 173 | 236

15. Primary Outcome: Number of Seroprotected Subjects Against the 3 Influenza Strains
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer ≥1:40.
Time Frame: At Day 21
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 50-64 Years Group | Fluarix 65+ Years Group | Fluarix 50+ Years Group
Number analyzed (Participants) | 171 | 307 | 478
Participants
  A/New Caledonia, Day 21 | 161 | 294 | 455
  A/Wisconsin, Day 21 | 144 | 280 | 424
  B/Malaysia, Day 21 | 155 | 290 | 445

16. Primary Outcome: Number of Seropositive Subjects for Each Influenza Strain
Description: A seropositive subject was defined as a vaccinated subject with antibody titer ≥1:10.
Time Frame: At Day 0 (PRE)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 50-64 Years Group | Fluarix 65+ Years Group | Fluarix 50+ Years Group
Number analyzed (Participants) | 171 | 307 | 478
Participants
  A/New Caledonia, PRE | 162 | 294 | 456
  A/Wisconsin, PRE | 102 | 209 | 311
  B/Malaysia, PRE | 132 | 277 | 409

17. Primary Outcome: Number of Seropositive Subjects for Each Influenza Strain
Description: A seropositive subject was defined as a vaccinated subject with an antibody titer ≥1:10.
Time Frame: At Day 21
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 50-64 Years Group | Fluarix 65+ Years Group | Fluarix 50+ Years Group
Number analyzed (Participants) | 171 | 307 | 478
Participants
  A/New Caledonia, Day 21 | 171 | 306 | 477
  A/Wisconsin, Day 21 | 167 | 304 | 471
  B/Malaysia, Day 21 | 168 | 306 | 474

18. Primary Outcome: Serum HI Antibody Titers for Each Influenza Strain
Description: Serum HI antibody titers were expressed as Geometric Mean Titers (GMTs).
Time Frame: At Day 0 (PRE)
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Fluarix 50-64 Years Group | Fluarix 65+ Years Group | Fluarix 50+ Years Group
Number analyzed (Participants) | 171 | 307 | 478
Titer
  A/New Caledonia, PRE | 40.5 [33.7 to 48.8] | 43.2 [38.3 to 48.7] | 42.2 [38.1 to 46.7]
  A/Wisconsin, PRE | 16.9 [13.8 to 20.8] | 21.5 [18.4 to 25.3] | 19.8 [17.4 to 22.4]
  B/Malaysia, PRE | 21.4 [18.0 to 25.4] | 38.8 [34.1 to 44.2] | 31.3 [28.2 to 34.9]

19. Primary Outcome: Serum HI Antibody Titers for Each Influenza Strain
Description: Serum HI antibody titers were expressed as Geometric Mean Titers (GMTs).
Time Frame: At Day 21
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Fluarix 50-64 Years Group | Fluarix 65+ Years Group | Fluarix 50+ Years Group
Number analyzed (Participants) | 171 | 307 | 478
Titer
  A/New Caledonia, Day 21 | 216.4 [180.8 to 259.0] | 142.9 [125.8 to 162.4] | 165.8 [149.2 to 184.2]
  A/Wisconsin, Day 21 | 156.7 [125.3 to 196.0] | 179.1 [154.0 to 208.4] | 170.8 [150.6 to 193.6]
  B/Malaysia, Day 21 | 149.9 [124.3 to 180.9] | 184.0 [161.9 to 209.2] | 171.0 [153.8 to 190.2]

ADVERSE EVENTS:
Time Frame: SAEs during the entire study period [from pre-season and up to the influenza surveillance period (from Month 0 up to Month 6)]
Description: Other (non-serious) Adverse Events were not collected
Arm/Group | Fluarix 50-64 Years Group | Fluarix 65+ Years Group
All-Cause Mortality (participants affected / at risk) | 2/1047 | 10/2007
Serious Adverse Events (participants affected / at risk) | 23/1047 | 105/2007
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluarix 50-64 Years Group (N=1047) | Fluarix 65+ Years Group (N=2007)
Myocardial infarction (Cardiac disorders) | 2 | 4
Angina pectoris (Cardiac disorders) | 0 | 5
Pneumonia (Infections and infestations) | 0 | 5
Atrial fibrillation (Cardiac disorders) | 0 | 4
Coronary artery disease (Cardiac disorders) | 0 | 4
Angina unstable (Cardiac disorders) | 1 | 2
Cardiac arrest (Cardiac disorders) | 1 | 2
Cerebrovascular accident (Nervous system disorders) | 1 | 2
Abdominal abscess (Infections and infestations) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Arrhythmia (Cardiac disorders) | 0 | 2
Chest pain (General disorders) | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1
Helicobacter gastritis (Infections and infestations) | 0 | 2
Hypoacusis (Ear and labyrinth disorders) | 1 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 1
Abscess (Infections and infestations) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Arterial occlusive disease (Vascular disorders) | 0 | 1
Arterial stenosis limb (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bleeding varicose vein (Vascular disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 0 | 1
Carotid artery stenosis (Vascular disorders) | 0 | 1
Chronic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Concussion (Nervous system disorders) | 0 | 1
Coronary artery occlusion (Vascular disorders) | 0 | 1
Death (General disorders) | 0 | 1
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 1
Femoral arterial stenosis (Vascular disorders) | 1 | 0
Femoral artery occlusion (Vascular disorders) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haematemesis (Vascular disorders) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Heart rate increased (Investigations) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Ischaemia (Vascular disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Organ failure (General disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Radial nerve palsy (Nervous system disorders) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal polyp (Gastrointestinal disorders) | 0 | 1
Retinal artery occlusion (Eye disorders) | 0 | 1
Retinitis (Eye disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Shock (Vascular disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Transient ischemic attack (Vascular disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
None reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.